CLINICAL TRIAL: NCT01361204
Title: Measurement of Stress Symptom in Students During Long-term Pharmacy Practices and Evaluation of Anti-stress Effect of Theanine Consumption on Students
Brief Title: Anti-stress Effect of Theanine on Students During Long-term Pharmacy Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Shizuoka (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT2011001
Record Dates: First submitted 2011-05-10; First posted 2011-05-26 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Students
Keywords: stress; students; pharmacy practice; theanine; pharmacy training
MeSH Terms: interventions — theanine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Theanine (Experimental): Experimental Comparator, theanine Taking 4 tablets of theanine two times daily for 16 days Placebo Comparator, sucrose Taking 4 tablets of sucrose two times daily for 16 days
  Interventions: Dietary Supplement: Theanine

INTERVENTIONS:
Dietary Supplement: Theanine — Taking 4 tablets of theanine two times daily for 16 days

SUMMARY:
Long-term practices in a hospital setting and community pharmacy might induce chronic stress in students. Alterations of salivary amylase activity will be measured in students during pharmacy practices as a marker of stress. Theanine is reported to have anti-stress effect on experimental animals under chronic stress and on humans under short-term stress. The purpose of this study is to measure stress symptoms in students during long-term pharmacy practices and to evaluate the efficacy of theanine in suppressing chronic stress, by measuring the salivary amylase activity.

DETAILED DESCRIPTION:
The investigators have found that theanine, an amino acid in green tea, has anti-stress and anti-aging effects using experimental animals. Mice, under chronic psychosocial stress, showed shortened longevity and brain dysfunction. However, when the mice ingested theanine, they showed normal longevity and brain function even though the mice were under psychosocial stress. These data showed that theanine has a significant anti-stress effect on mice. In addition, theanine has been reported to have an anti-stress effect on humans against short-term stress by measuring salivary amylase activity. However, the efficacy of theanine against chronic stress has not been examined. Long-term pharmacy practices might induce chronic stress in students. Based on this background, the investigators designed a randomized study to evaluate the clinical efficacy of theanine ingestion in suppressing chronic stress in students during long-term pharmacy practices.

ELIGIBILITY:
Inclusion Criteria:

* Students of pharmaceutical sciences in the fifth grade, nonsmoker
* Obtained written informed consent from the student before participation
* Possible to take tablets for 16 days
* Possible to check salivary amylase activity two times daily for 10 days

Exclusion Criteria:

* Taking tranquilizer(s)
* Smoker
* Diagnosed as inadequate to participate in the study by a doctor

Ages: 22 Months to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Alterations in salivary amylase activity in students with pharmacy practices | 10 days

SECONDARY OUTCOMES:
Numbers of students deteriorated physical condition | 10 days
Incidence of days of coming late or leaving early | 10 days
Alterations in sleeping hours from baseline | 10 days
Alterations in the response to a stress questionnaire from baseline | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Unno, Keiko, Principal Investigator — University of Shizuoka
Locations (1):
- University of Shizuoka, Shizuoka, Shizuoka, Japan